CLINICAL TRIAL: NCT05592626
Title: A Phase 1/2, First-in-Human, Open-Label, Dose Escalation and Expansion Study of STAR0602, a Selective T Cell Receptor (TCR) Targeting, Bifunctional Antibody-fusion Molecule, in Subjects With Unresectable, Locally Advanced, or Metastatic Solid Tumors That Are Antigen-rich (START-001)
Brief Title: A Study of a Selective T Cell Receptor (TCR) Targeting, Bifunctional Antibody-fusion Molecule STAR0602 in Participants With Advanced Solid Tumors
Acronym: START-001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marengo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-START-001
Record Dates: First submitted 2022-10-13; First posted 2022-10-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors; Genital Neoplasm, Female; Urogenital Neoplasms; Lung Neoplasm; Neoplasms by Site; Papillomavirus Infection; Epstein-Barr Virus Infections; Carcinoma; Neoplasms; Vulvar Neoplasms; Vulvar Diseases; Abdominal Neoplasm
Keywords: Advanced Solid Tumors; STAR0602; Intravenous; Antineoplastic Agents; T Cell Receptor-targeting; Bifunctional Antibody-Fusion; Specific T Cell Activator; Tumor Mutational Burden (TMB) High; Microsatellite Instability (MSI) High; Virally Associated Malignancies; Checkpoint Inhibitor Resistance; Immunotherapy; Immune Checkpoint Inhibitor Resistance; Head and Neck Cancer; Nasopharyngeal Cancer; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Biliary Cancer; Melanoma; Merkel Cell Carcinoma; Skin Squamous Cell Carcinoma; Skin Basal Cell Carcinoma; Endometrial Cancer; Colorectal Cancer; Small Bowel Cancer; Cervical Cancer; Gastrointestinal Neoplasms; Gastric Cancer; Esophageal Cancer; Bladder Cancer
MeSH Terms: conditions — Genital Neoplasms, Female; Urogenital Neoplasms; Lung Neoplasms; Neoplasms by Site; Papillomavirus Infections; Epstein-Barr Virus Infections; Carcinoma; Neoplasms; Vulvar Neoplasms; Vulvar Diseases; Abdominal Neoplasms; Microsatellite Instability; Head and Neck Neoplasms; Nasopharyngeal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Biliary Tract Neoplasms; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Basal Cell; Endometrial Neoplasms; Colorectal Neoplasms; Uterine Cervical Neoplasms; Gastrointestinal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1: Advanced Solid Tumors (Experimental): Dose Escalation; Intervention: Drug: STAR0602
  Interventions: Drug: STAR0602
- Phase 2: Advanced Solid Tumors (Experimental): Dose Expansion; Recommended Phase 2 Dose (RP2D) identified from Phase 1 will be used in Phase 2; Intervention: Drug: STAR0602
  Interventions: Drug: STAR0602

INTERVENTIONS:
Drug: STAR0602 — solution, intravenous infusion

SUMMARY:
This is an open label, multicenter, phase 1/2 study to assess the safety/tolerability and preliminary clinical activity of STAR0602 as a single agent administered intravenously in participants with advanced solid tumors that are antigen-rich.

DETAILED DESCRIPTION:
This Phase 1/2 study consists of two parts: Phase 1 Dose Escalation and Phase 2 Dose Expansion. In Phase 1 Dose Escalation, STAR0602 will be administered intravenously in participants with advanced solid tumors to assess safety/tolerability profile of STAR0602 and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of STAR0602. In Phase 2 Dose Expansion, STAR0602 at RP2D will be administered to participants with advanced, antigen-rich solid tumors to further evaluate safety and assess preliminary clinical activity of STAR0602. Clinical activity will be evaluated by objective tumor response rate (ORR), duration of response (DOR), disease control rate (DCR), and progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically confirmed solid tumors that are unresectable, locally advanced, or metastatic and for which standard curative therapies do not exist or are no longer effective or have intolerable toxicities. Subjects should not have received more than three lines of prior therapies for their advanced or metastatic diseases.
2. For Phase 1, participants must have one of the following solid tumors:

   1. High mutational burden (TMB-H)
   2. Microsatellite Instability (MSI-H)/DNA mismatch repair (dMMR)
   3. Virally associated tumors
3. For Phase 2, participants must have one of the following solid tumors:

   1. TMB-H
   2. MSI-H/dMMR
   3. CRC (both Ras wild type and mutant)
   4. Virally associated tumors
   5. Metastatic triple negative breast cancer
   6. Platinum-resistant epithelial ovarian cancer
   7. Metastatic castration-resistance prostate cancer
   8. Primary stage IV or recurrent non-small cell lung cancer
   9. Immunogenic solid tumors

   (Other tumor histologies may also be included in Phase 2 as additional data emerge to support their inclusion.)
4. Symptomatic central nervous system (CNS) metastases must have been treated, be asymptomatic for ≥ 14 days, and meet the following at the time of enrollment:

   * No concurrent treatment for CNS disease (e.g., surgery, radiation, corticosteroids > 10 mg prednisone/day or equivalent);
   * No concurrent leptomeningeal disease or cord compression.

Exclusion Criteria:

1. Participants with a history of known autoimmune disease with exceptions of:

   * Vitiligo;
   * Psoriasis, atopic dermatitis or other autoimmune skin condition not requiring systemic treatment;
   * History of Graves' disease, now euthyroid for > 4 weeks;
   * Hypothyroidism managed by thyroid replacement;
   * Alopecia;
   * Arthritis managed without systemic therapy beyond oral nonsteroidal anti-inflammatory drugs.
   * Adrenal insufficiency well controlled on replacement therapy.
2. Major surgery or traumatic injury within 8 weeks before first dose of study drug.
3. Unhealed wounds from surgery or injury.
4. Treatment with >10 mg per day of prednisone (or equivalent) or other immune-suppressive drugs within 7 days prior to the initiation of study drug. Exceptions may be made for patients who have had allergic reaction to iodinated contrast media. Steroids for topical, ophthalmic, inhaled, or nasal administration are allowed.
5. Clinically significant cardiovascular/vascular disease, gastrointestinal disorders, inflammatory processes, pulmonary compromises
6. Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of study drug.
7. Vaccination with any live virus vaccine within 4 weeks prior to the initiation of study drug administration. Inactivated annual influenza vaccination is allowed.
8. Participants who are known to be human immunodeficiency virus positive or hepatitis B or C positive and have uncontrolled disease.
9. Second primary invasive malignancy not in remission for ≥ 1 year. Exceptions include non-melanoma locally advanced skin cancer, cervical carcinoma in situ, localized prostate cancer (Gleason score ≤ 7), resected melanoma in situ, or any malignancy considered to be indolent and never required systemic therapy, with the exception of indolent lymphomas.
10. Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation).
11. Hepatic metastases unless adequately treated, either locally (e.g., by surgery, radiofrequency ablation, or chemoembolization) or systemically or both, and stable for 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose Escalation):Number of Participants with Dose-limiting Toxicities (DLTs) in Cycle 1 | Cycle 1 (Cycle length= 28 days)
Phase 1 and 2 (Dose Escalation and Expansion): Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 3 years
Phase 2 (Dose Expansion): Percentage of Participants with Overall Objective Tumor Responses (ORR) | Up to 3 years
  Complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Phase 1 and 2 (Dose Escalation and Expansion): Percentage of Participants with ORR | Up to 3 years
Phase 1 and 2 (Dose Escalation and Expansion): Duration of Responses (DOR) | Up to 3 years
Phase 1 and 2 (Dose Escalation and Expansion): Percentage of Participants with Disease Control (CR, PR, and Stable Disease) | Up to 3 years
Phase 2 (Dose Expansion): Progression Free Survival (PFS) | Up to 3 years
Phase 2 (Dose Expansion): Overall Survival (OS) | Up to 3 years
Phase 1 and 2 (Dose Escalation and Expansion): Maximum Observed Plasma Concentration (Cmax) for STAR0602 | Dose Escalation: Cycle 1 and Cycle 6 at predefined intervals up to 1 year; Dose Expansion: Cycle 1, Cycle 3, and Cycle 6 at predefined intervals up to 3 years (Cycle length= 28 days)
Phase 1 and 2 (Dose Escalation and Expansion): Time (Tmax) to Reach the Maximum Plasma Concentration (Cmax) for STAR0602 | Dose Escalation: Cycle 1 and Cycle 6 at predefined intervals up to 1 year; Dose Expansion: Cycle 1, Cycle 3, and Cycle 6 at predefined intervals up to 3 years (Cycle length= 28 days)
Phase 1 and 2 (Dose Escalation and Expansion): Area Under the Plasma Concentration (AUC) Versus Time Curve for STAR0602 | Dose Escalation: Cycle 1 and Cycle 6 at predefined intervals up to 1 year; Dose Expansion: Cycle 1, Cycle 3, and Cycle 6 at predefined intervals up to 3 years (Cycle length= 28 days)
Phase 1 and 2 (Dose Escalation and Expansion): Terminal Elimination Half-life (t1/2) for STAR0602 | Dose Escalation: Cycle 1 and Cycle 6 at predefined intervals up to 1 year; Dose Expansion: Cycle 1, Cycle 3, and Cycle 6 at predefined intervals up to 3 years (Cycle length= 28 days)
Phase 1 and 2 (Dose Escalation and Expansion): Apparent Total Body Clearance (CL) for STAR0602 | Dose Escalation: Cycle 1 and Cycle 6 at predefined intervals up to 1 year; Dose Expansion: Cycle 1, Cycle 3, and Cycle 6 at predefined intervals up to 3 years (Cycle length= 28 days)
Phase 1 and 2 (Dose Escalation and Expansion): Apparent Volume of Distribution (Vd) for STAR0602 | Dose Escalation: Cycle 1 and Cycle 6 at predefined intervals up to 1 year; Dose Expansion: Cycle 1, Cycle 3, and Cycle 6 at predefined intervals up to 3 years (Cycle length= 28 days)
Phase 1 and 2 (Dose Escalation and Expansion): Anti-drug Antibody (ADA) formation | Dose Escalation and Expansion: Day 1 of predetermined cycles up to 3 years (Cycle length= 28 days)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (18):
  - Loma Linda University Cancer Center, Loma Linda, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - AdventHealth Celebration, Celebration, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - The University of Kansas Cancer Center, Kansas City, Kansas
  - National Institutes of Health, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences, Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute Oncology Partners (SCRI-Nashville), Nashville, Tennessee
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - UT Health Mays Cancer Center, San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin- Madison, Madison, Wisconsin
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Research Institute of McGill University Health Centre, Montreal, Quebec
- France (5):
  - Hopsital Institut Curie, Paris, France
  - Oncopole Claudius Regaud IUCT, Toulouse, France
  - Institut Bergonié, Bordeaux
  - Centre Leon Berard, Lyon
  - Institute Gustave Roussy, Villejuif
- Spain (7):
  - Vall d'Hebron Institute of Oncology, Barcelona, Catalonia
  - Clinica Universidad de Navarra, San Blas-Canillejas, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid, Spain
  - NEXT Oncology Barcelona, Hospital Quirónsalud Barcelona, Barcelona
  - START Madrid FJD, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Instituto de Investigacion Sanitaria, INCLIVA, Valencia

IPD SHARING:
Plan to Share IPD: No